CLINICAL TRIAL: NCT01774162
Title: Endoscopic Ultrasound Guided Fine Needle Biopsy With a New Core Histology Needle Versus Conventional Fine Needle Aspiration.
Brief Title: EUS-guided Fine Needle Biopsy With a New Core Histology Needle Versus Conventional Fine Needle Aspiration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Christopher Teshima, Assistant Professor, University of Alberta
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00022017
Record Dates: First submitted 2013-01-18; First posted 2013-01-23 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Pancreas Adenocarcinoma; Pancreas Neoplasms; Gastrointestinal Stromal Tumor; Lymphoma
Keywords: Endoscopic Ultrasound; Fine needle aspiration; Fine needle biopsy; ProCore
MeSH Terms: conditions — Pancreatic Neoplasms; Gastrointestinal Stromal Tumors; Lymphoma | interventions — Biopsy, Fine-Needle; Cytological Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FNA for cytology (Active Comparator): Fine needle aspiration using conventional FNA for cytology
  Interventions: Device: Fine needle aspiration using conventional FNA for cytology
- FNB core biopsy for histology (Experimental): Fine needle biopsy using ProCore needle for histology.
  Interventions: Device: Fine needle biopsy using ProCore needle for histology.

INTERVENTIONS:
Device: Fine needle biopsy using ProCore needle for histology. — EUS-guided biopsy of each solid lesion using the EchoTip® ProCore™ ultrasound FNB needle for histology.
  Other Names: EchoTip® ProCore™ ultrasound FNB needle; Fine needle biopsy
  Arms: FNB core biopsy for histology
Device: Fine needle aspiration using conventional FNA for cytology — EUS-guided biopsy of each solid lesion using the EchoTip® Ultra™ FNA needle for cytology.
  Other Names: EchoTip® Ultra™ FNA needle; Fine needle aspiration
  Arms: FNA for cytology

SUMMARY:
Endoscopic ultrasound (EUS) is a well-established tool for the diagnosis and staging of many gastrointestinal conditions, including but not limited to, malignant and pre-malignant neoplasms of the pancreas, esophagus, rectum, and submucosal tumors developing along the gastrointestinal tract. EUS is the most sensitive test for the detection of focal lesions within the pancreas and is the most accurate method for diagnosing pancreas cancer. A biopsy method for tissue sampling via EUS called fine needle aspiration (FNA) was developed that enables a small needle to be passed into the lesion of interest under ultrasound guidance, obtaining cellular material for cytology. EUS-FNA is currently recommended for the diagnosis of cystic and solid mass lesions within and adjacent to the gastrointestinal tract. Yet in certain clinical circumstances, it is more desirable and sometimes necessary to obtain a core tissue biopsy for histology rather than the cellular material for cytology obtained with EUS-FNA. Furthermore, histology may generally increase the diagnostic yield of EUS-FNA compared to cytology. It is with these aims in mind that a new type of needle, the fine needle biopsy (EUS-FNB) device was developed to enable core tissue sampling. Since a comparison of these to methods has yet to be made, the aim of this study is to perform a direct comparison of the sampling adequacy and diagnostic yield of the new EUS-FNB needle with the conventional EUS-FNA needle.

DETAILED DESCRIPTION:
Background:

Endoscopic ultrasound (EUS) is a well-established tool for the diagnosis and staging of many gastrointestinal conditions, including but not limited to, malignant and pre-malignant neoplasms of the pancreas, esophagus, rectum, and submucosal tumors developing along the gastrointestinal tract. EUS provides endoscopic video imaging within the lumen of the gastrointestinal tract combined with ultrasound images via a transducer positioned at the tip of the endoscope. This diagnostic ability is enhanced by a biopsy method called fine needle aspiration (FNA). FNA via EUS (EUS-FNA) enables a small needle to be passed into a lesion of interest under ultrasound guidance, obtaining cellular material for cytology analysis. EUS-FNA is currently recommended for the confirmation of locally advanced pancreas adenocarcinoma, for the diagnosis of pancreatic cystic neoplasms and neuroendocrine tumors as well as autoimmune pancreatitis, for the characterization of submucosal tumors of the GI tract, and for the determination of malignant lymph node status in the staging of various cancers.

While EUS-FNA has an impressive technical success rate between 90-95%, the diagnostic accuracy is less robust for mass lesions, and in particular for pancreatic masses, for which the sensitivity and specificity is 75% and 100% respectively, translating into a negative predictive value of only 72%. And in the setting of chronic pancreatitis, a condition that is itself a major risk factor for the development of cancer and in which focal, non-malignant nodules often develop that may mimic tumors, the sensitivity of EUS-FNA may only be 54-74%. The diagnostic accuracy of EUS-FNA is of particular importance for pancreas adenocarcinoma and pancreatic neuroendocrine tumors because the 5-year survival rates are only 5% and 32% respectively. Thus, it is crucial that patients found to have a focal mass lesion have a reliable test that effectively excludes malignancy. Currently, EUS-FNA does not have the necessary negative predictive value in order to do so because the sensitivity of the test is too low. This means that a positive result on FNA confirms malignancy but that a negative result is unable to exclude it with confidence. This conundrum tends to leave the patient in the unfortunate position of having to often return for multiple investigations to perform repeat EUS-FNA when the clinical suspicion for a mass lesion remains high but the cytology result is thought to be falsely negative.

In order to overcome the current limitations of EUS-FNA cytology, the new EchoTip® ProCore™ fine needle biopsy (FNB) needle was developed in order obtain core tissue samples for both histology and cytology. This is important because histology is expected to increase the diagnostic yield of EUS-guided biopsy compared to cytology. In addition, in certain clinical circumstances it is more desirable and sometimes necessary to obtain a core tissue biopsy for histology rather than cellular material for cytology obtained with EUS-FNA.

In addition to the assessment of mass lesions in the pancreas, there are several other clinical areas in which the acquisition of core tissue samples for histology may prove superior to cytology from conventional EUS-FNA. For instance, EUS is part of the standard-of-care for the staging of esophageal cancer and histology may improve the sensitivity of EUS-biopsies for the determination of lymph node metastases. Also, although EUS is the preferred method for the work-up of submucosal lesions in the gastrointestinal tract, the value of EUS-FNA for differentiating the various subtypes of lesions is often limited, typically because FNA provides insufficient cellular material to reliably do so. Finally, it is clear that cytology from EUS-FNA is inadequate for the diagnosis of autoimmune pancreatitis and that a core biopsy sample for histology is needed. We expect the new EchoTip® ProCore™ FNB needle to potentially prove superior to FNA in all of these areas.

Study Objectives The purpose of this study is to determine if the new EchoTip® ProCore™ needle (FNB for histology) is superior to the current standard EchoTip® Ultra™ needle (FNA for cytology) for the diagnosis of focal, solid lesions for which biopsy sampling during EUS is clinically indicated. In particular, the objective is to compare the sampling adequacy of FNB with that of FNA for solid mass lesions within the pancreas, for submucosal lesions in the gastrointestinal tract and for the malignant status of lymph nodes as part of esophageal cancer staging. The sampling adequacy will be determined according to the ability of the pathologist to provide a definitive diagnostic interpretation based on the sample provided.

Study Design This is a prospective, comparative trial examining the use of the new EchoTip® ProCore™ FNB needle with the existing EchoTip® Ultra™ FNA needle stratified by lesion type (solid pancreas lesion, intra-abdominal mass, submucosal tumor, suspected metastatic lymph node). Both the FNB and FNA needle will be used in each lesion with randomization to needle type for first pass, alternating subsequent passes; thus each lesion will serve as its own internal control.

Methods Consecutive patients referred for EUS assessment of a solid lesion requiring FNA will be approached regarding study enrollment. Only those patients for whom EUS-FNA is clinically necessary will be selected. Consenting patients will undergo the standard EUS examination as indicated based on their lesion subtype, which will not differ from the EUS exam they would receive if they choose to not participate. Participating patients who have a lesion visualized during EUS that is technically amenable to FNA will then have their lesion biopsied by both FNB and FNA needles. The choice of needle size (19g or 22g) will be left to the clinical discretion of the endoscopist. However, the same needle size must be used for both the FNB and FNA needles.

Patients will be randomized to the type of needle used for the first pass into the lesion, with subsequent passes alternating between needle types. For the EchoTip® ProCore™ FNB needle, if a good sample is obtained (as assessed by the endoscopist performing the EUS examination) with the first pass, no further passes will be made. If the sample obtained with the first pass is considered likely insufficient or if no tissue was acquired, a second pass will then be performed. Regardless of what is obtained after the second needle pass, no additional passes will be made using the FNB. The core tissue obtained by the FNB needle will be placed in formalin and sent for histology analysis.

For the conventional EchoTip® Ultra™ FNA needle, a minimum of 2 passes will be performed. In cases in which a cytotechnologist is present, no feedback will be given to the endoscopist until after the 2nd pass. In cases where no cytotechnologist is present, up to 4 separate passes will be made, or fewer if the endoscopist is satisfied with the sample obtained. The sample obtained with the FNA needle will be placed on slides and also in cytology media (according to our standard clinical protocols).

The histology and cytology specimens will be sent to the pathology department at each site where the interpretation of samples will be done in the usual fashion as per standard clinical care. The pathologist will first describe the biopsy specimen in terms of the "adequacy of the sample for pathologist interpretation" - i.e. the ability of the pathologist to provide a definitive diagnostic interpretation based on the sample provided. Next, the pathologist will provide the diagnostic interpretation itself.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient 18 years or older
* Able to read and write English
* Undergoing EUS for the evaluation of: i) pancreas mass ii) intra-abdominal mass iii) suspected submucosal tumor iv) esophageal cancer staging v) other lymph node assessment

Exclusion Criteria:

* No detectable lesion
* lesion inaccessible to EUS guided biopsy
* Lesion determined to not require tissue sampling
* Pancreas lesion is predominantly cystic
* coagulopathy with a known clotting factor deficiency or an uncorrectable INR > 1.5, PTT > 40, platelet count < 50,000

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2011-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Sampling Adequacy | at time of procedure
  The ability of the pathologist to provide a definitive diagnostic interpretation (definitely positive, definitely negative or indeterminate reading) based on the tissue provided for a given lesion of interest.

SECONDARY OUTCOMES:
Sampling adequacy by lesion subtype | at time of procedure
  The sampling adequacy as defined in the primary outcome measure stratified by lesion subtype (pancreas, other intra-abdominal mass, liver mass, submucosal tumor, lymph node)
Diagnostic yield | at time of procedure
  The diagnosis obtained by FNA or FNB needle compared to the final diagnosis made by either FNA or FNB needle, subsequent surgery, or expert consensus at the end of the data collection period
Diagnostic yield by lesion subtype | at time of procedure
  The diagnosis obtained by the FNA or FNB needle compared to the final diagnosis obtained by either FNA or FNB needle, subsequent surgery or expert consensus regarding clinical diagnosis at the end of the data collection period.
Diagnostic agreement between FNA and FNB needles | at time of procedure
  The measure of agreement between diagnoses obtained by FNA and FNB needles for assessment of metastatic lymph nodes
Adverse events | at time of procedure
  Any adverse events including bleeding, fever, infection, pancreatitis, EUS-induced perforation, and sedation related complications occurring after both FNA and FNB biopsies.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher W Teshima, MD,FRCPC, Principal Investigator — University of Alberta
Locations (2):
- Canada (2):
  - Royal Alexandria Hospital, Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta

REFERENCES:
- [Background] Saftoiu A, Vilmann P. Role of endoscopic ultrasound in the diagnosis and staging of pancreatic cancer. J Clin Ultrasound. 2009 Jan;37(1):1-17. doi: 10.1002/jcu.20534. PMID 18932265
- [Background] Vilmann P, Jacobsen GK, Henriksen FW, Hancke S. Endoscopic ultrasonography with guided fine needle aspiration biopsy in pancreatic disease. Gastrointest Endosc. 1992 Mar-Apr;38(2):172-3. doi: 10.1016/s0016-5107(92)70385-x. No abstract available. PMID 1568614
- [Background] Maluf-Filho F, Dotti CM, Halwan B, Queiros AF, Kupski C, Chaves DM, Nakao FS, Kumar A. An evidence-based consensus statement on the role and application of endosonography in clinical practice. Endoscopy. 2009 Nov;41(11):979-87. doi: 10.1055/s-0029-1215192. Epub 2009 Oct 28. PMID 19866396
- [Background] Wiersema MJ, Vilmann P, Giovannini M, Chang KJ, Wiersema LM. Endosonography-guided fine-needle aspiration biopsy: diagnostic accuracy and complication assessment. Gastroenterology. 1997 Apr;112(4):1087-95. doi: 10.1016/s0016-5085(97)70164-1. PMID 9097990
- [Background] Eloubeidi MA, Tamhane A, Varadarajulu S, Wilcox CM. Frequency of major complications after EUS-guided FNA of solid pancreatic masses: a prospective evaluation. Gastrointest Endosc. 2006 Apr;63(4):622-9. doi: 10.1016/j.gie.2005.05.024. PMID 16564863
- [Background] Barawi M, Gottlieb K, Cunha B, Portis M, Gress F. A prospective evaluation of the incidence of bacteremia associated with EUS-guided fine-needle aspiration. Gastrointest Endosc. 2001 Feb;53(2):189-92. doi: 10.1067/mge.2001.108966. PMID 11174290
- [Background] Levy MJ, Norton ID, Wiersema MJ, Schwartz DA, Clain JE, Vazquez-Sequeiros E, Wilson WR, Zinsmeister AR, Jondal ML. Prospective risk assessment of bacteremia and other infectious complications in patients undergoing EUS-guided FNA. Gastrointest Endosc. 2003 May;57(6):672-8. doi: 10.1067/mge.2003.204. PMID 12709695
- [Background] Janssen J, Konig K, Knop-Hammad V, Johanns W, Greiner L. Frequency of bacteremia after linear EUS of the upper GI tract with and without FNA. Gastrointest Endosc. 2004 Mar;59(3):339-44. doi: 10.1016/s0016-5107(03)02707-x. PMID 14997128
- [Background] Smith EH. Complications of percutaneous abdominal fine-needle biopsy. Review. Radiology. 1991 Jan;178(1):253-8. doi: 10.1148/radiology.178.1.1984314.
- [Background] Micames C, Jowell PS, White R, Paulson E, Nelson R, Morse M, Hurwitz H, Pappas T, Tyler D, McGrath K. Lower frequency of peritoneal carcinomatosis in patients with pancreatic cancer diagnosed by EUS-guided FNA vs. percutaneous FNA. Gastrointest Endosc. 2003 Nov;58(5):690-5. doi: 10.1016/s0016-5107(03)02009-1. PMID 14595302
- [Background] Hirooka Y, Goto H, Itoh A, Hashimoto S, Niwa K, Ishikawa H, Okada N, Itoh T, Kawashima H. Case of intraductal papillary mucinous tumor in which endosonography-guided fine-needle aspiration biopsy caused dissemination. J Gastroenterol Hepatol. 2003 Nov;18(11):1323-4. doi: 10.1046/j.1440-1746.2003.03040.x. No abstract available. PMID 14535994
- [Background] Paquin SC, Gariepy G, Lepanto L, Bourdages R, Raymond G, Sahai AV. A first report of tumor seeding because of EUS-guided FNA of a pancreatic adenocarcinoma. Gastrointest Endosc. 2005 Apr;61(4):610-1. doi: 10.1016/s0016-5107(05)00082-9. No abstract available. PMID 15812422
- [Background] LeBlanc JK, Ciaccia D, Al-Assi MT, McGrath K, Imperiale T, Tao LC, Vallery S, DeWitt J, Sherman S, Collins E. Optimal number of EUS-guided fine needle passes needed to obtain a correct diagnosis. Gastrointest Endosc. 2004 Apr;59(4):475-81. doi: 10.1016/s0016-5107(03)02863-3. PMID 15044881
- [Background] Klapman JB, Logrono R, Dye CE, Waxman I. Clinical impact of on-site cytopathology interpretation on endoscopic ultrasound-guided fine needle aspiration. Am J Gastroenterol. 2003 Jun;98(6):1289-94. doi: 10.1111/j.1572-0241.2003.07472.x. PMID 12818271
- [Background] Erickson RA, Sayage-Rabie L, Beissner RS. Factors predicting the number of EUS-guided fine-needle passes for diagnosis of pancreatic malignancies. Gastrointest Endosc. 2000 Feb;51(2):184-90. doi: 10.1016/s0016-5107(00)70416-0. PMID 10650262
- [Background] Vilmann P, Saftoiu A. Endoscopic ultrasound-guided fine needle aspiration biopsy: equipment and technique. J Gastroenterol Hepatol. 2006 Nov;21(11):1646-55. doi: 10.1111/j.1440-1746.2006.04475.x. PMID 16984583
- [Background] Hartwig W, Schneider L, Diener MK, Bergmann F, Buchler MW, Werner J. Preoperative tissue diagnosis for tumours of the pancreas. Br J Surg. 2009 Jan;96(1):5-20. doi: 10.1002/bjs.6407. PMID 19016272
- [Background] Jemal A, Siegel R, Ward E, Hao Y, Xu J, Murray T, Thun MJ. Cancer statistics, 2008. CA Cancer J Clin. 2008 Mar-Apr;58(2):71-96. doi: 10.3322/CA.2007.0010. Epub 2008 Feb 20. PMID 18287387
- [Background] Levy MJ, Jondal ML, Clain J, Wiersema MJ. Preliminary experience with an EUS-guided trucut biopsy needle compared with EUS-guided FNA. Gastrointest Endosc. 2003 Jan;57(1):101-6. doi: 10.1067/mge.2003.49. PMID 12518144
- [Background] Levy MJ. Endoscopic ultrasound-guided trucut biopsy of the pancreas: prospects and problems. Pancreatology. 2007;7(2-3):163-6. doi: 10.1159/000104240. Epub 2007 Jun 21. PMID 17592229
- [Background] Larghi A, Verna EC, Stavropoulos SN, Rotterdam H, Lightdale CJ, Stevens PD. EUS-guided trucut needle biopsies in patients with solid pancreatic masses: a prospective study. Gastrointest Endosc. 2004 Feb;59(2):185-90. doi: 10.1016/s0016-5107(03)02538-0. PMID 14745390
- [Background] Varadarajulu S, Fraig M, Schmulewitz N, Roberts S, Wildi S, Hawes RH, Hoffman BJ, Wallace MB. Comparison of EUS-guided 19-gauge Trucut needle biopsy with EUS-guided fine-needle aspiration. Endoscopy. 2004 May;36(5):397-401. doi: 10.1055/s-2004-814316. PMID 15100946
- [Background] Itoi T, Itokawa F, Sofuni A, Nakamura K, Tsuchida A, Yamao K, Kawai T, Moriyasu F. Puncture of solid pancreatic tumors guided by endoscopic ultrasonography: a pilot study series comparing Trucut and 19-gauge and 22-gauge aspiration needles. Endoscopy. 2005 Apr;37(4):362-6. doi: 10.1055/s-2004-826156. PMID 15824948
- [Background] Polkowski M. Endosonographic staging of upper intestinal malignancy. Best Pract Res Clin Gastroenterol. 2009;23(5):649-61. doi: 10.1016/j.bpg.2009.05.002. PMID 19744630
- [Background] Puli SR, Reddy JB, Bechtold ML, Antillon D, Ibdah JA, Antillon MR. Staging accuracy of esophageal cancer by endoscopic ultrasound: a meta-analysis and systematic review. World J Gastroenterol. 2008 Mar 14;14(10):1479-90. doi: 10.3748/wjg.14.1479. PMID 18330935
- [Background] van Vliet EP, Heijenbrok-Kal MH, Hunink MG, Kuipers EJ, Siersema PD. Staging investigations for oesophageal cancer: a meta-analysis. Br J Cancer. 2008 Feb 12;98(3):547-57. doi: 10.1038/sj.bjc.6604200. Epub 2008 Jan 22. PMID 18212745
- [Background] Reed CE, Mishra G, Sahai AV, Hoffman BJ, Hawes RH. Esophageal cancer staging: improved accuracy by endoscopic ultrasound of celiac lymph nodes. Ann Thorac Surg. 1999 Feb;67(2):319-21; discussion 322. doi: 10.1016/s0003-4975(99)00031-4. PMID 10197647
- [Background] Philipper M, Hollerbach S, Gabbert HE, Heikaus S, Bocking A, Pomjanski N, Neuhaus H, Frieling T, Schumacher B. Prospective comparison of endoscopic ultrasound-guided fine-needle aspiration and surgical histology in upper gastrointestinal submucosal tumors. Endoscopy. 2010 Apr;42(4):300-5. doi: 10.1055/s-0029-1244006. Epub 2010 Mar 19. PMID 20306384
- [Background] Fernandez-Esparrach G, Sendino O, Sole M, Pellise M, Colomo L, Pardo A, Martinez-Palli G, Arguello L, Bordas JM, Llach J, Gines A. Endoscopic ultrasound-guided fine-needle aspiration and trucut biopsy in the diagnosis of gastric stromal tumors: a randomized crossover study. Endoscopy. 2010 Apr;42(4):292-9. doi: 10.1055/s-0029-1244074. Epub 2010 Mar 30. PMID 20354939
- [Background] Levy MJ, Wiersema MJ, Chari ST. Chronic pancreatitis: focal pancreatitis or cancer? Is there a role for FNA/biopsy? Autoimmune pancreatitis. Endoscopy. 2006 Jun;38 Suppl 1:S30-5. doi: 10.1055/s-2006-946648. No abstract available. PMID 16802220
- [Result] Chang KJ. Maximizing the yield of EUS-guided fine-needle aspiration. Gastrointest Endosc. 2002 Oct;56(4 Suppl):S28-34. doi: 10.1016/s0016-5107(02)70083-7. No abstract available. PMID 12297746